CLINICAL TRIAL: NCT03028337
Title: Single Versus Multifraction Salvage Spine Stereotactic Radiosurgery for Previously Irradiated Spinal Metastases: a Randomized Phase II Clinical Trial
Brief Title: Single Versus Multifraction Salvage Spine Stereotactic Radiosurgery for Previously Irradiated Spinal Metastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016-0728; NCI-2017-00606 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2017-01-19; First posted 2017-01-23 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Malignant Neoplasms of Eye Brain and Other Parts of Central Nervous System
Keywords: Malignant neoplasms of eye brain and other parts of central nervous system; Solid tumor malignancy; Radiographic evidence of spine metastasis; Spine radiosurgery; Radiation therapy; Radiotherapy; Questionnaires; Surveys; XRT
MeSH Terms: interventions — Radiotherapy; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spine Radiosurgery - 1 Dose (Experimental): Participants receive spine radiosurgery in a single large dose.
  Interventions: Radiation: Spine Radiosurgery; Behavioral: Questionnaires
- Spine Radiosurgery - 3 Doses (Active Comparator): Participants receive spine radiosurgery over 3 smaller doses.
  Interventions: Radiation: Spine Radiosurgery; Behavioral: Questionnaires

INTERVENTIONS:
Radiation: Spine Radiosurgery — Spine Radiosurgery - 1 Dose: For single fraction and multifraction arms, 0.01 cc of the cord allowed to receive 10 Gy and 14 Gy, respectively while 0.01 cc of the cauda equina allowed to receive 14 Gy and 18 Gy, respectively.
  Spine Radiosurgery - 3 Doses (3 days): The dose for the multifraction arm is 27 Gy in 3 fractions (9 Gy per fraction).
  Other Names: Radiotherapy; XRT
Behavioral: Questionnaires — Participants complete 3 questionnaires about any pain they may be having, quality-of-life, and any other symptoms. It should take about 10 minutes to complete these questionnaires.
  Questionnaires completed at Baseline and at Months 3,6,9,12,18, and 24 and then every 6 months after that during follow up.
  Other Names: Surveys

SUMMARY:
The goal of this clinical research study is to learn whether delivering spine radiosurgery in a single large dose is better than delivering spine radiosurgery over 3 smaller doses.

Researchers also want to learn about the effects of a single dose on participant's symptoms, pain, and quality-of-life.

DETAILED DESCRIPTION:
Study Groups:

Participant will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups. This is done because no one knows if one study group is better, the same, or worse than the other group.

* If participant is in Group 1, they will receive spine radiosurgery in a single large dose.
* If participant is in Group 2, they will receive spine radiosurgery over 3 smaller doses, which is standard.

Length of Study Participation:

Participant may continue taking part in the study as the doctor thinks it is in their best interest. Participant will no longer be able to take part if the disease gets worse, if intolerable side effects occur, or if they are unable to follow study directions.

Participation on the study will be over after participant's last follow-up visit.

Radiosurgery:

Participant will have spine radiosurgery in either 1 or 3 treatments as described above.

Participant will sign a separate consent for the surgery that explains the procedure and the risks.

Study Visits:

After surgery, at Months 3,6,9,12,18, and 24 and then every 6 months after that:

* Participant will have a physical exam, including a neurological exam (tests to check the functioning of their nerves, including tests of their strength and sensation.
* Participant will complete the same questionnaires they completed at the beginning of the study.
* Participant will have an MRI.

This is an investigational study. Delivering spine radiosurgery in a single large dose rather than over three smaller doses is considered investigational.

Up to 80 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must have histologic proof of solid tumor malignancy and radiographic evidence of spine metastasis
2. Age >/=18 years
3. Eastern Cooperative Oncology Group (ECOG) performance status </=2 (Karnofsky >/=60%)
4. Life expectancy of greater than 6 months
5. All patients must be able to lie supine
6. All patients must have no more than 3 contiguous vertebral body levels treated at a single site, and no more than 3 discontiguous vertebral body levels treated
7. All patients must have radiographic evidence of progression at a spinal site previously irradiated greater than 6 months prior to randomization. This includes indirect radiation exposure to spinal site.
8. All patients must have received prior conventional external-beam radiation therapy (cEBRT) to the site of interest to no more than a critical neural tissue dose equivalent dose (EQD)2/2 of 42 Gy in a single session or 50 Gy cumulative over multiple sessions and cauda equina dose EQD2/2 of 50 Gy in a single session or 60 Gy cumulative over multiple session. EQD2/2 is calculated as follows: EQD2/2= biologically effective dose (BED)/(1+d/alpha beta)) where BED=nd(1+d/(alpha beta)) and n=number of fractions, d=dose per fraction and alpha beta ratio of 2.
9. All patients must have a vertebral body site to be treated located from T1 to L5
10. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
11. All patients must sign informed consent verifying that they are aware of the investigational nature of this study in keeping with the rules and policies of MD Anderson Cancer Center. The only acceptable consent is the one approved by MD Anderson IRB.
12. Patients undergoing prior surgery or laser interstitial thermotherapy are allowed
13. Both men and women of all races and ethnic groups are eligible for this trial.

Exclusion Criteria:

1. Patients unable to undergo magnetic resonance imaging (MRI) of the spine
2. Prior radiation at the site of interest within 6 months
3. Prior history of radiation at the site of interest resulting in a critical neural tissue dose of EQD2/2 of >42 Gy in a single session
4. Patients unable to lie flat comfortably for 2 hours
5. Pregnancy status will be obtained at time of consent as is routine for all radiation patients. Pregnant women are excluded from this study because radiation has the potential for teratogenic or abortifacient effects
6. Patients with a histology of lymphoma and myeloma histologies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-01-18 (Actual); Primary Completion 2028-05-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Time to Local Failure Relative to Multi-Fraction Radiosurgery in Patients with Previously Irradiated Spinal Metastases | 12 months
  Local failure determined based on the surveillance MRI scan by study musculoskeletal radiologist.

SECONDARY OUTCOMES:
Pain Relief Relative to Multi-Fraction Radiosurgery in Patients with Previously Irradiated Spinal Metastases | 2 years
  Pain relief assessed by items on the Brief Pain Inventory (BPI) that measure severity, location, and degree of relief due to therapy by use of narcotic and non-narcotic pain medications and steroids. Patients experiencing a decrease of 2 points in the worst pain score for 2 consecutive assessment visits considered to have "partial pain relief". Complete pain relief defined as an average pain score of 0 for 2 consecutive assessment visits.

CONTACTS AND LOCATIONS:
Overall Officials: Amol J. Ghia, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org